CLINICAL TRIAL: NCT02018484
Title: Positioning of the Tibial Cut in Unicompartmental Medial Knee Replacement by Using Patient Specific Cutting Guides.
Acronym: PSI-PUC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2013-A01337-38
Record Dates: First submitted 2013-12-09; First posted 2013-12-23 (Estimated); Last update posted 2016-08-19 (Estimated); Status verified 2016-03

CONDITIONS: Knee Prosthesis
Keywords: Surgery / Knee / Replacement / MRI / Specific cutting guides
MeSH Terms: interventions — Arthroplasty, Replacement, Knee

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Patient specific cutting guides (Experimental): Unicompartmental knee replacement with patient specific cutting guides
  Interventions: Procedure: Unicompartmental Knee Replacement

INTERVENTIONS:
Procedure: Unicompartmental Knee Replacement

SUMMARY:
Unicompartmental knee replacements are performed to treat osteoarthritis or osteonecrosis of the knee especially when it affects only the medial femoro-tibial compartment. To place the prosthesis, bone removal is necessary. The orientations of the bony cuts directly influence the position of the different elements of the prosthesis and the limb alignment. It is known that good positioning of the prosthesis is the key of a good survival of the implants. To guide the blade of the saw, cutting guides are used. The position of these guides gives the final position of the cuts. At present, two main techniques are used to position the guides: the conventional one, not very costly but not very accurate, and the navigated procedure, which is more accurate but also more expensive and more invasive. Since few years, patient specific cutting guides are used in total knee replacement with encouraging results and more recently in uni compartmental knee replacement with no scientific proof of efficiency.

This study aims to validate the procedure of patient specific cutting guides.

DETAILED DESCRIPTION:
30 patients will be included in a mono centric, single-arm study with evaluation of the primary outcome by an independent expert comity. Each participant will have an MRI which will be sent to the society in charge of creating the patient specific cutting guides. The intervention will be performed using the patient specific cutting guides and in parallel, a station of navigation will be used to provide a safety control of the orientation of the cutting guide and to collect per operative data.

Evaluation visit is performed 6 months after surgery.

ELIGIBILITY:
Inclusion Criteria:

* patients aged 18 or older;
* indication of medial unicompartmental knee replacement (validated by the orthopedic surgeons staff) ;
* written informed consent.

Exclusion Criteria:

* MRI contraindication ;
* Absence of the main investigator or the associated scientist during the surgical procedure ;
* Adults under legal protective regimen or deprived of liberty.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2013-12; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Success rate in performing the tibial cut | Month 6
  Success is defined as a correct orientation of the tibial cut which has to be within patient's target value (± 2°) at 6 months in both the frontal and the sagittal plans.
  Failure of prosthesis implantation (defined by outranging patient's target value of more than 4º in the frontal or the sagittal plan or more than 3 mm on the cutting depth, controled by per operative navigated procedure) is considered as treatment failure.

SECONDARY OUTCOMES:
Success rate in conserving a residual varus. | Month 6
  Success is defined as a post-operative varus which does not exceed the patient's target value ± 3°, while respecting a 1° minimal varus.
Variations of other orientation parameters of the tibial cut and limb alignment at the different times of the procedure (per and post operative) . | Per-operative, and Month 6

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Christophe Lambotte, MD, Principal Investigator — Rennes University Hospital; Bruno Laviolle, MD, PhD, Study Chair — CIC INSERM 0203 CHU de RENNES
Locations (1):
- Chu Rennes, Rennes, France